CLINICAL TRIAL: NCT06433622
Title: Platelet Transfusion and Repeat Thromboelastography With Platelet Mapping (TEG-PM) in Patients With Severe Traumatic Brain Injuries (TBI) on Antiplatelet Therapy
Brief Title: Platelet Transfusion and Repeat TEG-PM in Patients With Severe TBI on Antiplatelet Therapy (Repeat TEG-PM)
Status: Enrolling by invitation | Type: Observational
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Principal Investigator, Lindsey Perea, Trauma and Acute Care Surgeon, Lancaster General Hospital
Other Study IDs: 2023-47
Record Dates: First submitted 2024-04-30; First posted 2024-05-30 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Traumatic Intracranial Hemorrhage
MeSH Terms: conditions — Intracranial Hemorrhage, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Repeat TEG-PM: Will receive a repeat TEG-PM after platelet transfusion based on inclusion criteria.
  Interventions: Diagnostic Test: Repeat Thromboelastography with Platelet Mapping
- No Repeat TEG-PM: Not eligible to be consented; will proceed with normal course of treatment.

INTERVENTIONS:
Diagnostic Test: Repeat Thromboelastography with Platelet Mapping — Thromboelastography (TEG) is an assay used by many medical professionals to assess coagulopathy, predict outcomes, and guide treatment. Although TEG does not assess platelet function very well, a TEG with platelet mapping (TEG-PM) assay assesses platelet functioning by measuring the percent of arachidonic acid (AA) and adenosine diphosphate (ADP) that are inhibited in the patient's blood.
  Groups: Repeat TEG-PM

SUMMARY:
The aim of this study is to see if administering platelets (cells in our blood that stop or prevent bleeding) results in improved platelet function and slows/stops the progression of a head bleed for patients who have a traumatic head bleed and are on antiplatelet therapy (medications that stop blood cells from forming a blood clot) prior to admission.

DETAILED DESCRIPTION:
This study aims to determine if platelet function has improved following platelet transfusion by prospectively performing repeat thromboelastographic with platelet mapping (TEG-PM) assays on all patients consented and enrolled in the study. This study will also examine the rate of progression or stability of ICH on repeat head CT following platelet administration and will aid in the determination of a potential association between repeat CT head findings and the repeat TEG-PM results.

ELIGIBILITY:
Inclusion Criteria for Interventional Portion of Study:

* Patients ≥ 18 years of age who present with TICH meeting Brain Injury Guidelines (BIG) 2 or 3 head bleed criteria
* Currently on antiplatelet medication on admission
* Must have taken this antiplatelet medication within the past 48 hours prior to presentation
* Patients who have AA and/or ADP inhibition of 70% or greater and Maximum Amplitude (MA) <50 will then receive a platelet transfusion and a repeat TEG-PM 1hr after transfusion

Exclusion Criteria for Interventional Portion of Study:

* Under 18 years of age
* Have a known bleeding diatheses
* Current therapeutic anticoagulation use
* Do not know the time of their last antiplatelet medication dose
* Patients or their proxy who are unable to provide consent
* Patients with concomitant long bone fractures or solid organ injuries

Inclusion Criteria for Retrospective Portion of Study:

• Patients with a TICH who are 18 years of age or older

Exclusion Criteria for Retrospective Portion of Study:

* Abbreviated Injury Scale (AIS) >1 in body regions other than head because of concomitant long bone fracture or solid organ injury
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targeted population includes patients ≥ 18 years of age who present to Penn Medicine Lancaster General Health with TICH. Selection of subjects is based on all adult patients presenting with TICH that are admitted to Lancaster General Health Trauma Center.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Repeat TEG | 1 hour after platelets given
  Rate of reversed pathway inhibition on repeat thromboelastography with platelet mapping (TEG-PM) when platelets are administered to TICH patients who are on antiplatelet therapy prior to admission.
Repeat Head CT | From the time of interventional platelet administration until the time of patient discharge from their index admission, assessed up to 100 weeks.
  Number of patients with improved platelet function on repeat TEG-PM and stability of TICH on subsequent CT scan.

SECONDARY OUTCOMES:
Need for Neurosurgical Intervention | During index admission for traumatic intracranial hemorrhage (TICH), assessed through study completion, an average of 2 years.
  Determine the efficacy of platelet transfusion among this patient cohort by measuring need for neurosurgical intervention after second CT scan (ie: the failure of non-operative management)
Discharge Status | From the time of interventional platelet administration until the time of patient discharge from their index admission assessed through study completion, an average of 2 years.
  Determine the efficacy of platelet transfusion among this patient cohort by reviewing discharge status.

OTHER OUTCOMES:
Mortality | During index admission for traumatic intracranial hemorrhage (TICH), assessed through study completion, an average of 2 years.
  Determine the efficacy of platelet transfusion among this patient cohort by measuring mortality rate.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Perea, DO, Principal Investigator — Penn Medicine Lancaster General Health
Locations (1):
- Penn Medicine Lancaster General Health, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Traumatic brain injury: time to end the silence. Lancet Neurol. 2010 Apr;9(4):331. doi: 10.1016/S1474-4422(10)70069-7. No abstract available. PMID 20298955
- [Background] Li L, Geraghty OC, Mehta Z, Rothwell PM; Oxford Vascular Study. Age-specific risks, severity, time course, and outcome of bleeding on long-term antiplatelet treatment after vascular events: a population-based cohort study. Lancet. 2017 Jul 29;390(10093):490-499. doi: 10.1016/S0140-6736(17)30770-5. Epub 2017 Jun 13. PMID 28622955
- [Background] Pace WD. Daily Low-Dose Aspirin, Diabetes, and Age-Still Looking for a Balance. JAMA Netw Open. 2021 Jun 1;4(6):e2112875. doi: 10.1001/jamanetworkopen.2021.12875. No abstract available. PMID 34152422
- [Background] Alter SM, Mazer BA, Solano JJ, Shih RD, Hughes MJ, Clayton LM, Greaves SW, Trinh NQ, Hughes PG. Antiplatelet therapy is associated with a high rate of intracranial hemorrhage in patients with head injuries. Trauma Surg Acute Care Open. 2020 Nov 25;5(1):e000520. doi: 10.1136/tsaco-2020-000520. eCollection 2020. PMID 33294625
- [Background] van den Brand CL, Tolido T, Rambach AH, Hunink MG, Patka P, Jellema K. Systematic Review and Meta-Analysis: Is Pre-Injury Antiplatelet Therapy Associated with Traumatic Intracranial Hemorrhage? J Neurotrauma. 2017 Jan 1;34(1):1-7. doi: 10.1089/neu.2015.4393. Epub 2016 May 9. PMID 26979949
- [Background] Svedung Wettervik T, Lenell S, Enblad P, Lewen A. Pre-injury antithrombotic agents predict intracranial hemorrhagic progression, but not worse clinical outcome in severe traumatic brain injury. Acta Neurochir (Wien). 2021 May;163(5):1403-1413. doi: 10.1007/s00701-021-04816-0. Epub 2021 Mar 26. PMID 33770261
- [Background] Peck KA, Calvo RY, Schechter MS, Sise CB, Kahl JE, Shackford MC, Shackford SR, Sise MJ, Blaskiewicz DJ. The impact of preinjury anticoagulants and prescription antiplatelet agents on outcomes in older patients with traumatic brain injury. J Trauma Acute Care Surg. 2014 Feb;76(2):431-6. doi: 10.1097/TA.0000000000000107. PMID 24458049
- [Background] Fabbri A, Servadei F, Marchesini G, Bronzoni C, Montesi D, Arietta L; Societa Italiana di Medicina d'Emergenza Urgenza Study Group. Antiplatelet therapy and the outcome of subjects with intracranial injury: the Italian SIMEU study. Crit Care. 2013 Mar 21;17(2):R53. doi: 10.1186/cc12575. PMID 23514619
- [Background] Joseph B, Pandit V, Aziz H, Kulvatunyou N, Hashmi A, Tang A, O'Keeffe T, Wynne J, Vercruysse G, Friese RS, Rhee P. Clinical outcomes in traumatic brain injury patients on preinjury clopidogrel: a prospective analysis. J Trauma Acute Care Surg. 2014 Mar;76(3):817-20. doi: 10.1097/TA.0b013e3182aafcf0. PMID 24553554
- [Background] Van Ornam J, Pruitt P, Borczuk P. Is repeat head CT necessary in patients with mild traumatic intracranial hemorrhage. Am J Emerg Med. 2019 Sep;37(9):1694-1698. doi: 10.1016/j.ajem.2018.12.012. Epub 2018 Dec 10. PMID 30559018
- [Background] Shammassian BH, Ronald A, Smith A, Sajatovic M, Mangat HS, Kelly ML. Viscoelastic Hemostatic Assays and Outcomes in Traumatic Brain Injury: A Systematic Literature Review. World Neurosurg. 2022 Mar;159:221-236.e4. doi: 10.1016/j.wneu.2021.10.180. Epub 2021 Nov 27. PMID 34844010
- [Background] Fleming K, Redfern RE, March RL, Bobulski N, Kuehne M, Chen JT, Moront M. TEG-Directed Transfusion in Complex Cardiac Surgery: Impact on Blood Product Usage. J Extra Corpor Technol. 2017 Dec;49(4):283-290. PMID 29302119
- [Background] Fan D, Ouyang Z, Ying Y, Huang S, Tao P, Pan X, Lu S, Pan Q. Thromboelastography for the Prevention of Perioperative Venous Thromboembolism in Orthopedics. Clin Appl Thromb Hemost. 2022 Jan-Dec;28:10760296221077975. doi: 10.1177/10760296221077975. PMID 35379018
- [Background] Rao A, Lin A, Hilliard C, Fu R, Lennox T, Barbosa R, Schreiber M, Rowell S. The Utility of Thromboelastography for Predicting The Risk of Progression of Intracranial Hemorrhage in Traumatic Brain Injury Patients. Neurosurgery. 2017 Sep 1;64(CN_suppl_1):182-187. doi: 10.1093/neuros/nyx210. No abstract available. PMID 28899039
- [Background] Kay AB, Morris DS, Collingridge DS, Majercik S. Platelet dysfunction on thromboelastogram is associated with severity of blunt traumatic brain injury. Am J Surg. 2019 Dec;218(6):1134-1137. doi: 10.1016/j.amjsurg.2019.09.024. Epub 2019 Sep 23. PMID 31575420
- [Background] Davis PK, Musunuru H, Walsh M, Cassady R, Yount R, Losiniecki A, Moore EE, Wohlauer MV, Howard J, Ploplis VA, Castellino FJ, Thomas SG. Platelet dysfunction is an early marker for traumatic brain injury-induced coagulopathy. Neurocrit Care. 2013 Apr;18(2):201-8. doi: 10.1007/s12028-012-9745-6. PMID 22847397
- [Background] Nekludov M, Bellander BM, Blomback M, Wallen HN. Platelet dysfunction in patients with severe traumatic brain injury. J Neurotrauma. 2007 Nov;24(11):1699-706. doi: 10.1089/neu.2007.0322. PMID 18001200
- [Background] Daley MJ, Enright Z, Nguyen J, Ali S, Clark A, Aydelotte JD, Teixeira PG, Coopwood TB, Brown CV. Adenosine diphosphate platelet dysfunction on thromboelastogram is independently associated with increased morality in traumatic brain injury. Eur J Trauma Emerg Surg. 2017 Feb;43(1):105-111. doi: 10.1007/s00068-016-0643-z. Epub 2016 Feb 18. PMID 26888580
- [Background] Cannon JW, Dias JD, Kumar MA, Walsh M, Thomas SG, Cotton BA, Schuster JM, Evans SL, Schreiber MA, Adam EH, Zacharowski K, Hartmann J, Schochl H, Kaplan LJ. Use of Thromboelastography in the Evaluation and Management of Patients With Traumatic Brain Injury: A Systematic Review and Meta-Analysis. Crit Care Explor. 2021 Sep 14;3(9):e0526. doi: 10.1097/CCE.0000000000000526. eCollection 2021 Sep. PMID 34549189
- [Background] Lee J, Kim JK, Kim JH, Dunuu T, Park SH, Park SJ, Kang JY, Choi RK, Hyon MS. Recovery time of platelet function after aspirin withdrawal. Curr Ther Res Clin Exp. 2014 Mar 25;76:26-31. doi: 10.1016/j.curtheres.2014.02.002. eCollection 2014 Dec. PMID 25031665
- [Background] Glass NE, Riccardi J, Horng H, Kacprzynski G, Sifri Z. Platelet dysfunction in patients with traumatic intracranial hemorrhage: Do desmopressin and platelet therapy help or harm? Am J Surg. 2022 Jan;223(1):131-136. doi: 10.1016/j.amjsurg.2021.07.050. Epub 2021 Aug 3. PMID 34446216
- [Background] Wolff C, Muakkassa F, Marley R, El-Khatib A, Docherty C, Muakkassa L, Stephen H, Salvator A. Routine platelet transfusion in patients with traumatic intracranial hemorrhage taking antiplatelet medication: Is it warranted? Can J Surg. 2022 Mar 15;65(2):E206-E211. doi: 10.1503/cjs.018120. Print 2022 Mar-Apr. PMID 35292527
- [Background] Miles MVP, Hicks RC, Parmer H, Brown C, Edwards A, Stewart K, Gao L, Maxwell R. Traumatic brain injury patients with platelet inhibition receiving platelet transfusion demonstrate decreased need for neurosurgical intervention and decreased mortality. J Trauma Acute Care Surg. 2022 Apr 1;92(4):701-707. doi: 10.1097/TA.0000000000003516. PMID 35320155
- [Background] Jehan F, Zeeshan M, Kulvatunyou N, Khan M, O'Keeffe T, Tang A, Gries L, Joseph B. Is There a Need for Platelet Transfusion After Traumatic Brain Injury in Patients on P2Y12 Inhibitors? J Surg Res. 2019 Apr;236:224-229. doi: 10.1016/j.jss.2018.11.050. Epub 2018 Dec 20. PMID 30694760
- [Background] Lokhandwala AM, Asmar S, Khurrum M, Chehab M, Bible L, Castanon L, Ditillo M, Joseph B. Platelet Transfusion After Traumatic Intracranial Hemorrhage in Patients on Antiplatelet Agents. J Surg Res. 2021 Jan;257:239-245. doi: 10.1016/j.jss.2020.07.076. Epub 2020 Aug 27. PMID 32862051
- [Background] Spiess BD. Platelet transfusions: the science behind safety, risks and appropriate applications. Best Pract Res Clin Anaesthesiol. 2010 Mar;24(1):65-83. doi: 10.1016/j.bpa.2009.11.001. PMID 20402171
- [Background] Joseph B, Pandit V, Sadoun M, Larkins CG, Kulvatunyou N, Tang A, Mino M, Friese RS, Rhee P. A prospective evaluation of platelet function in patients on antiplatelet therapy with traumatic intracranial hemorrhage. J Trauma Acute Care Surg. 2013 Dec;75(6):990-4. doi: 10.1097/TA.0b013e3182a96591. PMID 24256671
- [Background] Holzmacher JL, Reynolds C, Patel M, Maluso P, Holland S, Gamsky N, Moore H, Acquista E, Carrick M, Amdur R, Hancock H, Metzler M, Dunn J, Sarani B. Platelet transfusion does not improve outcomes in patients with brain injury on antiplatelet therapy. Brain Inj. 2018;32(3):325-330. doi: 10.1080/02699052.2018.1425804. Epub 2018 Jan 17. PMID 29341793
- See also: Get the facts about TBI. Centers for Disease Control and Prevention. — https://www.cdc.gov/traumatic-brain-injury/data-research/facts-stats/?CDC_AAref_Val=https://www.cdc.gov/traumaticbraininjury/get_the_facts.html
- See also: Facts about falls. Centers for Disease Control and Prevention. — https://www.cdc.gov/falls/data-research/facts-stats/?CDC_AAref_Val=https://www.cdc.gov/falls/facts.html
- See also: TBI data. Centers for Disease Control and Prevention. — https://www.cdc.gov/traumatic-brain-injury/data-research/?CDC_AAref_Val=https://www.cdc.gov/traumaticbraininjury/data/index.html
- See also: United Zion Retirement Community. Why Retire to Lititz in Lancaster County? Retirement Advice. February 11, 2019. — http://www.uzrc.org/blog/retirement-advice/retire-to-lititz/
- See also: Word Population Review. Lancaster County, Pennsylvania Population 2022. World Population Review. 2022. — https://worldpopulationreview.com/us-counties/pa/lancaster-county-population